CLINICAL TRIAL: NCT07288957
Title: A Phase 1, First-in-Human, Multicenter, Open-Label Study of ABSK131 to Assess Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy in Patients With MTAP-Deficient Advanced/Metastatic Solid Tumors
Brief Title: A Early Study of ABSK131 in Patients With Advanced/Metastatic Solid Tumors
Acronym: ABSK131-101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABSK131-101
Record Dates: First submitted 2025-11-25; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors (Phase 1)
Keywords: ABSK131; MTAP; PRMT5

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Escalation and expansion part (Experimental): No more than 86 patients are anticipated to be enrolled in the escalation part. No more than 180 patients will be enrolled in the expansion part
  Interventions: Drug: ABSK131

INTERVENTIONS:
Drug: ABSK131 — In the escalation part，patients will first orally receive a single dose of ABSK131 on D-2, followed by a two-day run-in period to assess the PK profile of single-dose ABSK131 administration. Thereafter, patients will continuously receive ABSK131 once daily (QD).
  In the expansion part， patients will orally receive ABSK131 at the recommended dose for expansion (RDE)

SUMMARY:
This is a first-in-human (FIH), multicenter, non-randomized, openlabel, phase 1 study of ABSK131 in patients with MTAP-Deficient Advanced/Metastatic Solid Tumors to evaluate the safety, tolerability, PK, and preliminary antitumor efficacy.

DETAILED DESCRIPTION:
The study will be started with a dose escalation part of ABSK131 administered in repeated 21-day cycles in patients with MTAP-Deficient Advanced/Metastatic Solid Tumors. The expansion part of oral ABSK131 at the recommended dose of expansion (RDE) will be followed to evaluate safety, tolerability, and preliminary antitumor activity among patients with MTAP-Deficient Advanced/Metastatic Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients should understand, sign, and date the written informed consent form before screening.
* 2. Male or female aged 18 years or older.
* 3. Patients with histologically or cytologically confirmed metastatic or locally advanced solid tumor; have received and progressed, are refractory or are intolerant to standard therapy or lack of standard therapy for the particular tumor type.
* 4. Patients with homozygous deletion of MTAP gene based on central testing or sponsor-accepted local report (depending on the availability of regional genetic testing), or with MTAP expression loss in the tumor based on the central testing.
* 5. Patients should provide archival tumor sample or undergo tumor biopsy at baseline if archival sample is not available or inadequate.
* 6. Backfill cohorts and expansion cohorts: Patients with 1 of the following cancers and have received no more than 3 prior lines of therapy。1)NSCLC；2) Pancreatic cancer；3)Esophageal cancer；4)Gastric cancer；5)Mesotheliomas.

Food effect: a. Be able to eat a standardized high-fat meal within 30 minutes. b. Without primary GI tumors or metastasis.

* 7. Patients must have at least one measurable target lesion according to RECIST v1.1.
* 8. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* 9. Life expectancy ≥3 months.
* 10.Adequate organ function and bone marrow function as indicated by the screening assessments performed within 14 days prior to the first dose of study drug.
* 11.Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to the first dose.
* 12.Non-surgically sterilized male or female patients of childbearing potential must agree to use highly effective methods of birth control from signing the informed consent to approximately 6 months after the last dose of study drug. A condom is also required to be used by vasectomized men to prevent delivery of the drug via seminal fluid.

Exclusion Criteria:

* 1. Known allergy or hypersensitivity to any component of ABSK131.
* 2. Prior treatment with a PRMT5 or MAT2A inhibitor therapy.
* 3. Another active primary malignancy.
* 4. Unable to swallow capsules or malabsorption syndrome, disease significantly affecting GI function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction, or current evidence of GI disease that present with diarrhea. If any of these conditions exist, the sites' staff should discuss with the sponsor to determine patient eligibility.
* 5. Any of the situation within the specified time frame prior to the first administration of study drug.
* 6. Prior toxicities from chemotherapy, radiotherapy, and other anti-cancer therapies, including immunotherapy that have not regressed to Grade ≤ 1 severity (CTCAE v5.0) with the exception of which eligibility criteria allows, or alopecia, vitiligo, hypothyroidism stable on hormone replacement, or Grade 2 peripheral neurotoxicity.
* 7. Potent strong inhibitors or inducers of CYP3A family within 2 weeks before the first dose of study treatment (3 weeks for St John's Wort); consumption of grapefruit juice, grapefruit hybrids, pomegranates, starfruits, pomelos, seville oranges or juice products within 3 days prior to the first dose of study treatment.
* 8. Proton pump inhibitors, such as omeprazole, lansoprazole, dexlansoprazole, or pantoprazole within 7 days before the first dose of study treatment.
* 9. Imaging (CT or MRI) showed tumor invasion of large blood vessels (such as aorta, pulmonary artery, pulmonary vein, vena cava, etc.) or risk of bleeding (such as esophageal and gastric varices).
* 10.Have current spinal cord compression (symptomatic or asymptomatic and detected by radiographic imaging) or leptomeningeal disease (symptomatic or asymptomatic) or symptomatic unstable brain metastases. Patients with a history of brain metastases have been treated and are stable ≥ 28 days may be enrolled. Patients with no steroid use for at least 2 weeks prior to the time of enrollment are permitted.
* 11.Impaired cardiac function or clinically significant cardiac disease.
* 12.Known acquired immunodeficiency syndrome (AIDS)-related illness, or positive test for HIV 1/2 antibody.
* 13.Exclusion of hepatitis infection.
* 14.Patients with ascites or pleural effusion, or pericardial effusion which is refractory/uncontrolled, or requiring the intervention within 2 weeks prior to the first dose.
* 15.Confirmed or suspected ILD/pneumonitis or history of (non-infectious) ILD/pneumonitis that required oral or IV steroids or supplemental oxygen.
* 16.Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test within 7 days prior to the start of study drug.
* 17.Vaccination with a live, attenuated vaccine within 4 weeks prior to the first dose of study treatment except for administration of inactivate vaccines .
* 18.Has had an allogenic tissue/solid organ transplant.
* 19.Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* 20.Any other clinically significant comorbidities, such as uncontrolled pulmonary disease, active infection, or any other condition, which in the judgment of investigators, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | from Run-in to Day21
  Dose-limiting toxicities
AEs | The date of signing the informed consent form until 30 days (including Day 30) after the last dose of study drug, assessed up to 30 months.
  Adverse events
AESIs | he date of signing the informed consent form until 30 days (including Day 30) after the last dose of study drug, assessed up to 30 months.
  Adverse events of special interest (AESIs)
SAEs | The date of signing the informed consent form until 30 days (including Day 30) after the last dose of study drug, assessed up to 30 months
  Serious adverse events (SAEs)

SECONDARY OUTCOMES:
Cmax | From date of enrollment（Run-） until the date of end of treatment visit, assessed up to 30 months
  Maximum observed concentration
AUC | From date of enrollment（R） until the date of end of treatment visit, assessed up to 30 months
  area under the concentration-time curve
t1/2 | From date of enrollment（Run-in） until the date of end of treatment visit, assessed up to 30 months
  elimination half-life
CL/F | From date of enrollment（Run-in） until the date of end of treatment visit, assessed up to 30 months
  apparent oral clearance
tmax | From date of enrollment（R） until the date of end of treatment visit, assessed up to 30 months
  time to maximum observed concentration
ORR | From date of enrollment（R）until the date of disease progression, start of new anticancer treatment, death, withdrawal of consent of study, lost to follow up or end of study, whichever comes first，assessed up to 30 months
  Objective response rate
DOR | From date of enrollment（R）until the date of disease progression, start of new anticancer treatment, death, withdrawal of consent of study, lost to follow up or end of study, whichever comes first，assessed up to 30 months
  Duration of response
PFS | From date of enrollment（R）until the date of disease progression, start of new anticancer treatment, death, withdrawal of consent of study, lost to follow up or end of study, whichever comes first，assessed up to 30 months
  Progression-free survival
DCR | From date of enrollment（R）until the date of disease progression, start of new anticancer treatment, death, withdrawal of consent of study, lost to follow up or end of study, whichever comes first，assessed up to 30 months
  Disease control rate
OS | From date of enrollment（Run-in）until the date of death, withdrawal of consent of study, lost to follow up or end of study, whichever comes first，assessed up to 60 months
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No